CLINICAL TRIAL: NCT00814073
Title: Randomized, Placebo-controlled, Phase 3 Study to Compare Efficacy and Safety of Masitinib at 6 mg/kg/Day to Placebo in Treatment of Patients With Smouldering Systemic, Indolent Systemic or Cutaneous Mastocytosis With Handicap
Brief Title: Masitinib in Severe Indolent or Smoldering Systemic Mastocytosis
Acronym: AB06006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB06006
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: Mastocytosis with handicap; Mastocytosis; Mast cell; Mast cell infiltration; Skin; Bone marrow; Pruritus; Flushes; c-kit; c-kit mutation; Wild Type; Mutation Asp-816-Val(D816V); Indolent systemic mastocytosis; smoldering systemic mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis; Pruritus; Blushing; Piebaldism | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib & BSC (Experimental): Masitinib (6 mg/kg/day) administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC)
  Interventions: Drug: Masitinib; Other: Best Supportive Care
- Placebo & BSC (Placebo Comparator): Matching placebo administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC)
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: Masitinib — Masitinib 6 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib & BSC
Drug: Placebo — Matching placebo
  Arms: Placebo & BSC
Other: Best Supportive Care — Optimal concomitant symptomatic treatments. Includes: H1- and H2-antihistamines, proton pump inhibitors (PPI), sodium cromoglicate, antidepressants, leukotriene antagonists, interferon-alpha, 2-CdA, and corticosteroids.

SUMMARY:
The objective of this study is to compare the safety and efficacy of masitinib (AB1010) to placebo in patients with mastocytosis with handicap.

DETAILED DESCRIPTION:
This was a prospective, multicenter, randomized, placebo-controlled, parallel-group, phase 3 study, conducted in 15 countries, evaluating the efficacy and safety of masitinib (6 mg/kg/day administered orally in two daily intakes over 24-weeks with a double-blind extension period possible) for the treatment of indolent systemic mastocytosis, smoldering mastocytosis or cutaneous mastocytosis, in patients with mast cells mediator release symptoms that are refractory to conventional symptomatic treatment.

A study protocol amendment restricted enrolment to patients with severe indolent and smoldering systemic mastocytosis. The objective of this phase 3 study was therefore to evaluate masitinib efficacy and safety in severe systemic mastocytosis patients, with or without D816V mutation of c-Kit. The primary objective of the phase 3 study was to detect a statistically significant difference between masitinib (plus optimal concomitant symptomatic treatments) and placebo (plus optimal concomitant symptomatic treatments) in cumulative response on four severe symptoms, referred to also as handicaps.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with one of the following documented mastocytosis as per WHO classification: Smouldering Systemic Mastocytosis, Severe Indolent Mastocytosis
2. Patient with documented mastocytosis and evaluable disease based upon histological criteria: typical infiltrates of mast cells in a multifocal or diffuse pattern in skin and/or bone marrow biopsy
3. Patient with documented treatment failure of his/her handicap(s) with at least one of the following therapy used at optimized dose: Anti H1, Anti H2, Proton pump inhibitor, Osteoclast inhibitor, Cromoglycate Sodium, Antileukotriene
4. Handicapped status defined as at least two of the following handicaps, including at least one among pruritus, flushes, depression and fatigue: pruritus score ≥ 9, number of flushes per week ≥ 8, Hamilton rating scale for depression (HAMD-17) score ≥ 19, number of stools per day ≥ 4, number of mictions per day ≥ 8, Fatigue Impact Scale total score (asthenia) ≥ 75
5. Patients with OPA ≥ 2 (moderate to intolerable general handicap)
6. ECOG ≤ 2
7. Patient with adequate organ function

Exclusion Criteria:

1. Patient with one of the following mastocytosis: Cutaneous Mastocytosis, Not documented Smouldering Systemic Mastocytosis or Indolent Systemic Mastocytosis, Systemic Mastocytosis with an Associated clonal Hematologic Non Mast cell lineage Disease (SM-AHNMD), Mast cell leukemia (MCL), Aggressive systemic mastocytosis (ASM)
2. Previous treatment with any Tyrosine Kinase Inhibitor
3. Patient with recent cardiac history of: Acute coronary syndrome, Acute heart failure, Significant ventricular arrhythmia; patient with cardiac failure class III or IV; Syncope without known aetiology within 3 months, uncontrolled severe hypertension.
4. Patient with any condition that the physician judges could be detrimental to subjects participating in this study; including any clinically important deviations from normal clinical laboratory values or concurrent medical events Previous treatment
5. Change in the symptomatic treatment of mastocytosis or administration of any new treatment of mastocytosis within 4 weeks prior to baseline
6. Treatment with any investigational agent within 4 weeks prior to baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cumulative response (4R75%) | 24 weeks
  The prospectively declared primary endpoint (4R75%) was cumulative response in at least one of four severe baseline symptoms of mast cell mediator release (pruritus, flushes, depression, or asthenia). Response was defined as a 75% improvement from baseline for any of these four symptoms. Cumulative response was defined as the number of actual responses between weeks 8 and 24, divided by the total number of possible responses over the same treatment period (ie, with five scheduled visits, each patient had a maximum of five to 20 possible responses depending on the number of severe baseline symptoms).

SECONDARY OUTCOMES:
Cumulative response (3R75%) | 24 weeks
  Cumulative response in at least one of three severe baseline symptoms (pruritus, flushes, or depression)
Cumulative response (2R75%) | 24 weeks
  Cumulative response in at least one of three severe baseline symptoms (pruritus or flushes)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, MD, PhD, Principal Investigator — Hôpital Necker, Paris, France
Locations (24):
- United States (2):
  - UC Davis Health System , Department of Dermatology, Sacramento, California
  - MD Anderson Cancer Centre, Houston, Texas
- France (22):
  - CHU d'Amiens, Amiens
  - Hôpital Avicenne, Bobigny
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Claude Huriez, Lille
  - CHU Dupuytren, Limoges
  - Hôpital Ambroise Paré, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Central, Nancy
  - CHU Hôtel Dieu, Nantes
  - Hôpital l'Archet II, Nice
  - Hôpital Necker, Paris
  - Hôpital Tenon, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Milétrie, Poitiers
  - CHU Hôpital Sud, Rennes
  - CHU de Saint-Etienne, Saint-Etienne
  - Hôpital Purpan, Toulouse
  - Hôpital Bretonneau, Tours
  - Hôpital des Hauts Clos, Troyes

REFERENCES:
- [Background] Arock M. A new therapeutic advance for symptomatic systemic mastocytosis? Lancet. 2017 Feb 11;389(10069):576-578. doi: 10.1016/S0140-6736(16)31655-5. Epub 2017 Jan 7. No abstract available. PMID 28069280
- [Result] Lortholary O, Chandesris MO, Bulai Livideanu C, Paul C, Guillet G, Jassem E, Niedoszytko M, Barete S, Verstovsek S, Grattan C, Damaj G, Canioni D, Fraitag S, Lhermitte L, Georgin Lavialle S, Frenzel L, Afrin LB, Hanssens K, Agopian J, Gaillard R, Kinet JP, Auclair C, Mansfield C, Moussy A, Dubreuil P, Hermine O. Masitinib for treatment of severely symptomatic indolent systemic mastocytosis: a randomised, placebo-controlled, phase 3 study. Lancet. 2017 Feb 11;389(10069):612-620. doi: 10.1016/S0140-6736(16)31403-9. Epub 2017 Jan 7. PMID 28069279
- See also: Publication of results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5985971/